CLINICAL TRIAL: NCT04074434
Title: Study Watch Atrial Fibrillation (AF) Detection Investigation
Status: Completed | Type: Observational
Sponsor: Verily Life Sciences LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 100145
Record Dates: First submitted 2019-08-22; First posted 2019-08-30 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All Participants
  Interventions: Device: Study Watch

INTERVENTIONS:
Device: Study Watch — Study Watch is a miniaturized physiological data monitoring and data collection device for continuous recording of physiological and environmental data

SUMMARY:
This is a prospective, non-randomized study to refine the Study Watch's algorithm for AF detection within both persistent and paroxysmal AF subjects. The study will also collect data from an FDA-cleared wearable ECG sensor.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Able to read and speak English
* Able and willing to sign written Informed Consent
* Interest in participating in the study
* Subjects with a known history of AF (including persistent or paroxysmal AF)
* Without significant limitation in ability to participate in the study, in the opinion of the investigator.

Exclusion Criteria:

* Currently in a paced rhythm
* Known severe allergy to nickel or metal jewelry
* Known allergic reaction to adhesives or hydrogels or with family history of adhesive skin allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a known history of AF (including persistent or paroxysmal AF)
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Estimate of the accuracy of algorithm based PPG irregular rhythm detection in a study population with a history of paroxysmal or persistent atrial fibrillation (AF) | At least 60 minutes
  Sensitivity estimate for PPG irregular rhythm detection vs. a multi-lead Holter ECG rhythm
PPG- and ECG-based continuous AF-detection algorithms on Study Watch in a free-living (home) setting by comparing the Study Watch data with an FDA-cleared wearable ECG sensor data. | 14 days
  Number of AF events identified from FDA-cleared ECG Device

SECONDARY OUTCOMES:
Estimate of the accuracy of algorithm based PPG irregular rhythm detection in a study population with a history of paroxysmal or persistent atrial fibrillation (AF) | At least 60 minutes
  Predictive value estimate for PPG irregular rhythm detection vs. a multi-lead Holter ECG rhythm
Spontaneously-reported participant usability feedback for Study Watch and its ECG feature in a free-living (home) setting with the target AF population. | 14 days
  Qualitative listing of participant-reported feedback

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego Cardiac Center, San Diego, California, United States